CLINICAL TRIAL: NCT07049536
Title: Investigation of Physical Fitness Parameters of Allogeneic Stem Cell Transplant Recipients
Brief Title: Physical Fitness of Allogeneic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Asst. Prof., Istinye University
Other Study IDs: 24-03
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: physical fitness; stem cell transplantation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transplantation Group: Adult patients who underwent hematopoietic stem cell transplantation
  Interventions: Other: Assessment Group
- Control Group: Healthy adults
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Assessment Group — Allogeneic Stem Cell Transplant recipients will be evaluated with a supervisor physiotherapist for 2 days between the time they are admitted to the stem cell transplantation unit.
  Groups: Transplantation Group
Other: Control Group — Adult healthy group with similar sociodemographic characteristics to the evaluation group.
  Groups: Control Group

SUMMARY:
Hematopoietic stem cell transplantation is a treatment used to restore blood cell function in diseases of myeloid and lymphoid origin, which can be malignant or non-malignant. There are two types: autologous transplantation, which uses the patient's own stem cells, and allogeneic transplantation, which uses stem cells from a donor after a high-dose chemotherapy and radiotherapy preparation. This process can lead to complications such as immune reactions, infections, and organ toxicity, affecting the cardiovascular, musculoskeletal, and nervous systems. These complications often reduce physical activity, muscle strength, lung function, and quality of life.

Before transplantation, it is important to assess patients' comorbidities, functional status, and physical fitness to evaluate their ability to tolerate treatment and risk of complications. Low exercise tolerance and impaired physical function are linked to poorer outcomes. Objective tests of physical function provide valuable information about health status. Pre-transplant muscle strength and cardiopulmonary fitness influence post-transplant recovery, so comprehensive assessments are necessary.

Physiotherapy and rehabilitation support patients by preparing them for treatment, maintaining health during therapy, improving physical function after treatment, and enhancing quality of life in palliative care. Exercise improves functional capacity, quality of life, and daily activities, but symptoms like fatigue, pain, breathlessness, and muscle weakness, as well as other barriers, may limit participation.

Physical fitness is the body's ability to perform daily activities efficiently. Reduced fitness leads to frailty and decreased function, which are associated with increased treatment toxicity and mortality. Although the importance of physical fitness before transplantation is recognized, data from objective measurements are limited. Common pre-transplant assessments include lung function tests, walking tests, handgrip strength, and mobility tests.

This study aims to compare the health-related physical fitness of individuals undergoing allogeneic hematopoietic stem cell transplantation with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving treatment in the Adult Bone Marrow Transplantation Unit
* Between 18 and 65 years of age
* Undergoing standard medical treatment including immunosuppressants, antibiotics, and other medications
* Clinically stable, able to walk, and cooperative
* No history of orthopedic, neurological, or cardiac disorders

Exclusion Criteria:

* Presence of cognitive impairments
* Orthopedic or neurological diseases that may affect the evaluation of physical fitness tests
* Presence of facial palsy
* Severe visual impairment or visual field defects
* Acute bleeding, hemoglobin level ≤ 8 g/dL, and platelet count ≤ 10,000/mm³

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 30 individuals will be included in the study, consisting of 15 adult patients who have undergone hematopoietic stem cell transplantation and meet the inclusion criteria from the Adult Bone Marrow Transplantation Unit, forming the research group, and 15 healthy individuals forming the control group. RPatients and healthy controls will be matched based on age and gender.The study will commence following Ethics Committee approval and will be conducted in accordance with the principles of the Declaration of Helsinki. Informed consent will be obtained from all participants included in the study.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in One Second | 4 weeks
  The volume of air that can be forcefully exhaled during the first second of a forced breath.
Forced Vital Capacity | 4 weeks
  The total volume of air that can be forcibly exhaled after taking the deepest breath possible.
Forced Expiratory Volume in One Second to Forced Vital Capacity Ratio | 4 weeks
  The percentage ratio of the volume of air exhaled in the first second to the total volume exhaled during the forced vital capacity test.
Peak Expiratory Flow | 4 weeks
  The maximum speed of expiration during a forced breath.
Physical Activity Level: | 4 weeks
  The level of physical activity will be assessed using the Turkish version of the short form of the International Physical Activity Questionnaire. This questionnaire was developed to measure health-related physical activity in populations and is both comprehensive and concise. It provides information on the time spent sitting, walking, and engaging in moderate and vigorous intensity physical activities.
  The total score is calculated by multiplying the duration and frequency of the physical activities reported. The energy expenditure associated with physical activities is expressed in metabolic equivalent-minute scores. Based on the scoring, the questionnaire categorizes individuals into three physical activity levels: inactive, moderately active, and active.
  The administration of the questionnaire can be conducted in two different formats: on paper or via a digital screen interface.
Six-Minute Walk Test | 4 weeks
  Functional exercise capacity will be evaluated using the Six-Minute Walk Test in accordance with the criteria of the American Thoracic Society and the European Respiratory Society. In this test, the individual is instructed to walk as fast as possible back and forth between two cones placed 30 meters apart in a straight corridor.
  Standardized encouragement phrases will be used throughout the test to motivate the participant. Vital signs will be assessed before and after the test, as well as during the recovery period. The total distance walked during the six-minute period will be recorded in meters, and the average walking speed will be calculated in meters per minute.
Postural Assessment: | 4 weeks
  The Posture Analysis Form developed by Corbin will be used for the assessment of postural alignment. The evaluation will be conducted through visual observation from both lateral and posterior views. The presence and severity of postural deviations will be assessed. Each item in the form is scored based on the severity of the deviation as follows:
  0 = none, 1 = mild, 2 = moderate, 3 = severe. The total score will be used to classify the individual's overall postural status.
Sit and Reach Test | 4 weeks
  Sit and Reach Test reflects lower body flexibility. In this test, the patient will be seated in front of a box with dimensions of 35 cm length, 45 cm width, 32 cm height, and after leaning his bare feet on the inner surface of the box, patient will try to move the bar on the plate as far as patient can with both hands, the value at the last point will be recorded in cm.
Assessment of Respiratory Muscle Strength | 4 weeks
  Respiratory muscle strength will be evaluated by measuring maximum inspiratory mouth pressure and maximum expiratory mouth pressure using a portable electronic mouth pressure measurement device. Results will be recorded in cmH₂O.
  Maximum inspiratory mouth pressure is defined as the pressure generated in the mouth during maximal inspiration against an occluded airway. For this measurement, participants will first perform a maximal expiration, after which the airway will be closed with a valve, and the participant will be asked to perform a maximal inspiration sustained for 1-3 seconds.
  maximum expiratory mouth pressure refers to the pressure generated in the mouth during maximal expiration against a closed airway. For maximum expiratory mouth pressure measurement, after a maximal inspiration, the participant will be instructed to exhale maximally against the occluded airway for 1-3 seconds.
Assessment of Peripheral Muscle Strength | 4 weeks
  Peripheral muscle strength will be assessed for the following muscle groups: shoulder abductors, shoulder flexors, elbow flexors and extensors for the upper extremity; and hip flexors and knee extensors for the lower extremity. Measurements will be performed using a portable manual muscle strength testing device (Model 01165, Lafayette, Indiana, United States of America).
Grip strength | 4 weeks
  Grip strength will be assessed using a Jamar Hydraulic Hand Dynamometer (Jamar, Nottinghamshire, United Kingdom). Measurements will be performed in a seated position with the elbow flexed at 90 degrees and the wrist in a neutral position.
  Measurements for both right and left sides will be repeated three times, and the best value obtained will be recorded in kilograms.
30-Second Sit-to-Stand Test | 4 weeks
  In this test, the participant is asked to sit down and stand up from a standard chair as many times as possible within 30 seconds, without using their arms. The number of full stands completed within the allotted time is recorded. This test provides functional information about lower extremity muscle strength.
Flamingo Balance Test | 4 weeks
  In this test, the participant is asked to stand barefoot in a flamingo-like position and maintain balance for as long as possible. The participant balances on one leg, while the other leg is flexed so that the foot touches the opposite knee. A stopwatch is started upon command. Each time balance is lost, the timer is paused, and restarted once balance is regained. The total number of balance losses within 1 minute is recorded. If the participant loses balance more than 15 times within the first 30 seconds, the test is terminated and scored as zero.
Semmes-Weinstein Monofilament Test | 4 weeks
  This test is performed to assess light touch and pressure sensations. The assessment tool consists of a series of monofilaments with varying thickness and diameters. These monofilaments apply graded forces ranging from 0.086 grams to 448 grams. The evaluation begins with the smallest monofilament and proceeds sequentially to thicker ones. The test is stopped, and the value is recorded, when the smallest monofilament perceived by the participant is identified. The monofilaments are applied from the first to the fifth finger, moving from distal to proximal regions, on both anterior and posterior surfaces of the hand.
Quality of Life Assessment | 4 weeks
  Quality of life, including physical and mental health components, will be assessed using the Short Form 36 Health Survey Questionnaire. The Short Form 36 is a 36-item self-report questionnaire that evaluates eight dimensions of health: physical functioning, role limitations due to physical health, role limitations due to emotional problems, social functioning, bodily pain, mental health, vitality, and general health perceptions. In addition to individual subscale scores, two summary scores-physical component summary and mental component summary-are calculated by combining the relevant subscales.

SECONDARY OUTCOMES:
Height | 4 weeks
  The vertical distance from the top of the head to the heels of the individual. It will be measured in centimeters.
Weight | 4 weeks
  The mass of the individual's body in relation to gravity. It will be expressed in kilograms.
Demographic data and physical characteristics | 4 weeks
  The sociodemographic status of the participants will be recorded with an evaluation form prepared by the researchers. Information on age, gender, dominant side, exercise habits will be questioned. Data regarding diagnosis, disease stage, and treatments (chemotherapy/radiotherapy) will be obtained from the hospital medical record information processing system.Participants' privacy will be respected throughout the study, and no photographs will be taken.
Waist Circumference Measurement | 4 weeks
  To assess waist circumference, participants will be asked to stand upright with arms relaxed at their sides and feet together. A non-elastic measuring tape will be held horizontally and parallel to the ground, and the measurement will be taken from the narrowest part of the torso. The measurement will be performed twice, and the average of the two values will be recorded in centimeters.
Hip Circumference Measurement: | 4 weeks
  Hip circumference will be measured with the participant standing with feet together. A non-elastic measuring tape will be placed horizontally at the widest part of the buttocks. The measurement will be taken twice, and the average of the two readings will be recorded in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided